CLINICAL TRIAL: NCT02702492
Title: A Phase 1 Open-Label Study of the Safety, Tolerability and Efficacy of KPT-9274, a Dual Inhibitor of PAK4 and NAMPT, in Patients With Advanced Solid Malignancies or Non-Hodgkin's Lymphoma
Brief Title: PAK4 and NAMPT in Patients With Solid Malignancies or NHL (PANAMA)
Acronym: PANAMA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCP-9274-901
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumors; NHL
Keywords: PAK4; KPT-9274; Karyopharm; NHL; Solid Tumors; NAMPT; Melanoma
MeSH Terms: conditions — Melanoma | interventions — KPT-9274; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Part A: KPT-9274 10mg (Experimental): Participants received a 10 milligrams (mg) of oral tablets of KPT-9274 three times a week every other day during each 28 day cycle.
  Interventions: Drug: KPT-9274
- Part A: KPT-9274 20mg (Experimental): Participants received a 20mg of oral tablets of KPT-9274 three times a week every other day during each 28 day cycle.
  Interventions: Drug: KPT-9274
- Part A: KPT-9274 30mg (Experimental): Participants received a 30mg of oral tablets of KPT-9274 three times a week every other day during each 28 day cycle.
  Interventions: Drug: KPT-9274
- Part A: KPT-9274 40mg (Experimental): Participants received a 40mg of oral tablets of KPT-9274 three times a week every other day during each 28 day cycle.
  Interventions: Drug: KPT-9274
- Part A: KPT-9274 40mg BIW (Experimental): Participants received KPT-9274 40mg of oral tablet biweekly (BIW) during each 28-day cycle.
  Interventions: Drug: KPT-9274
- Part B: KPT-9274 30mg + Niacin 500mg (Experimental): Participants received KPT-9274 30mg of oral tablet along with a starting dose of 500mg niacin extended release (ER) orally three times a week every other day during each 28-day cycle.
  Interventions: Drug: KPT-9274; Drug: Niacin ER
- Part B: KPT-9274 40mg + Niacin 500mg (Experimental): Participants received KPT-9274 40mg of oral tablet along with a starting dose of 500mg niacin ER orally three times a week every other day during each 28-day cycle.
  Interventions: Drug: KPT-9274; Drug: Niacin ER
- Part B: KPT-9274 60mg + Niacin 500mg (Experimental): Participants received KPT-9274 60mg of oral tablet along with a starting dose of 500mg niacin ER orally three times a week every other day during each 28-day cycle.
  Interventions: Drug: KPT-9274; Drug: Niacin ER
- Part B: KPT-9274 80mg + Niacin 500mg (Experimental): Participants received KPT-9274 80mg of oral tablet along with a starting dose of 500mg niacin ER orally three times a week every other day during each 28-day cycle.
  Interventions: Drug: KPT-9274; Drug: Niacin ER
- Part B: KPT-9274 100mg + Niacin 500mg (Experimental): Participants received KPT-9274 100mg of oral tablet along with a starting dose of 500mg niacin ER orally three times a week every other day during each 28-day cycle.
  Interventions: Drug: KPT-9274; Drug: Niacin ER
- Part C: KPT-9274 20mg + Nivolumab 480mg (Experimental): Participants received KPT-9274 20mg of oral tablet three times a week every other day during each 28-day cycle along with 480mg of nivolumab intravenous infusion on Day 1 of each cycle (once every 4-week cycle).
  Interventions: Drug: KPT-9274; Drug: Nivolumab
- Part C: KPT-9274 30mg + Nivolumab 480mg (Experimental): Participants received KPT-9274 30mg of oral tablet three times a week every other day during each 28-day cycle along with 480mg of nivolumab intravenous infusion on Day 1 of each cycle (once every 4-week cycle).
  Interventions: Drug: KPT-9274; Drug: Nivolumab
- Part C: KPT-9274 40mg + Nivolumab 480mg (Experimental): Participants received KPT-9274 40mg of oral tablet three times a week every other day during each 28-day cycle along with 480mg of nivolumab intravenous infusion on Day 1 of each cycle (once every 4-week cycle).
  Interventions: Drug: KPT-9274; Drug: Nivolumab

INTERVENTIONS:
Drug: KPT-9274
Drug: Niacin ER
  Arms: Part B: KPT-9274 100mg + Niacin 500mg; Part B: KPT-9274 30mg + Niacin 500mg; Part B: KPT-9274 40mg + Niacin 500mg; Part B: KPT-9274 60mg + Niacin 500mg; Part B: KPT-9274 80mg + Niacin 500mg
Drug: Nivolumab
  Other Names: Opdivo®
  Arms: Part C: KPT-9274 20mg + Nivolumab 480mg; Part C: KPT-9274 30mg + Nivolumab 480mg; Part C: KPT-9274 40mg + Nivolumab 480mg

SUMMARY:
This study will evaluate the safety, tolerability, and efficacy of oral KPT-9274 for the treatment of patients with advanced solid malignancies or non-Hodgkin's lymphoma (NHL).

DETAILED DESCRIPTION:
This is a first-in-human, multi-center, open-label clinical study with separate Dose Escalation and Expansion Phases to assess preliminary safety, tolerability, and efficacy of KPT-9274, a dual inhibitor of PAK4 and NAMPT, in patients with advanced solid malignancies (including sarcoma, colon, lung, melanoma, etc.) or NHL for which all standard therapeutic options considered useful by the investigator have been exhausted.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria to be eligible to enroll in the Part C of this study.

1. Should have unresectable advanced, recurrent or metastatic melanoma and must have objective and measurable melanoma by RECIST 1.1 after disease progression on a prior anti-PD-1 or anti-PD-L1 therapy.
2. ECOG performance status of ≤ 2.
3. Life expectancy of ≥ 3 months.
4. Adequate hepatic function:

   * Total bilirubin < 1.5 times the ULN (except participants with Gilbert's syndrome [hereditary indirect hyperbilirubinemia] who must have a total bilirubin of ≤ 3 times ULN),
   * AST and ALT ≤ 2.5 times ULN (except participants with known liver involvement of their advanced solid malignancy who must have an AST and ALT ≤ 5.0 times ULN).
5. Adequate renal function:

   * Estimated creatinine clearance of ≥ 60 mL/min, calculated using the formula of Cockroft and Gault (140-Age) Mass (kg)/(72 creatinine mg/dL); multiply by 0.85 if female.
6. Adequate hematopoietic function:

   * Total WBC count ≥ 1500/mm³, ANC ≥ 1000/mm³, Hb ≥ 10.0 g/dL, platelet count ≥ 100,000/mm³

Exclusion Criteria:

Participants meeting any of the following exclusion criteria are not eligible to enroll in this study.

1. ≤ 2 weeks since the last prior therapeutic regimen for melanoma. Palliative steroids for disease related symptoms < 7 days prior to C1D1, unless physiologic doses of steroids are used.
2. Have not recovered or stabilized (Gr 1 or to their baseline for non-hematologic toxicities, ≤ Gr 2 or to their baseline for hematologic toxicities) from toxicities related to their previous treatment except for alopecia.
3. Untreated CNS disease or leptomeningeal involvement are excluded. Participants without active brain or leptomeningeal metastases after prior treatment with local therapies are eligible provided that the treatment had been done ≥ 2 weeks prior to enrollment.
4. Active infection with completion of therapeutic antibiotics, antivirals, or antifungals within one week prior to C1D1. Prophylactic antibiotics, antivirals or antifungals are permitted.
5. Significantly diseased or obstructed gastrointestinal tract or uncontrolled vomiting or diarrhea that could interfere with the absorption of KPT-9274.
6. Active peptic ulcer disease or other active gastrointestinal bleeds.
7. Requiring treatment with corticosteroids at doses higher than substitute therapy (> 10 mg prednisone), are unstable with substitute hormonal therapy, or are deemed to be likely to re-occur by the treating physician when administered nivolumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-01-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - UCLA Health, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Georgetown University, Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Mayo Clinic Rochester, Rochester, Minnesota
  - NYU-Laura & Isaac Perlmutter Cancer Center, New York, New York
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Han W, Yang Y, Yu F, Li Q, Liu A, Xu W, Li J, Xue X. Design, synthesis and anticancer activity evaluation of 4-(3-1H-indazolyl)amino quinazoline derivatives as PAK4 inhibitors. Bioorg Med Chem. 2023 Nov 15;95:117501. doi: 10.1016/j.bmc.2023.117501. Epub 2023 Oct 13. PMID 37864885
- [Derived] Mpilla GB, Uddin MH, Al-Hallak MN, Aboukameel A, Li Y, Kim SH, Beydoun R, Dyson G, Baloglu E, Senapedis WT, Landesman Y, Wagner KU, Viola NT, El-Rayes BF, Philip PA, Mohammad RM, Azmi AS. PAK4-NAMPT Dual Inhibition Sensitizes Pancreatic Neuroendocrine Tumors to Everolimus. Mol Cancer Ther. 2021 Oct;20(10):1836-1845. doi: 10.1158/1535-7163.MCT-20-1105. Epub 2021 Jul 12. PMID 34253597
- [Derived] Aboukameel A, Muqbil I, Senapedis W, Baloglu E, Landesman Y, Shacham S, Kauffman M, Philip PA, Mohammad RM, Azmi AS. Novel p21-Activated Kinase 4 (PAK4) Allosteric Modulators Overcome Drug Resistance and Stemness in Pancreatic Ductal Adenocarcinoma. Mol Cancer Ther. 2017 Jan;16(1):76-87. doi: 10.1158/1535-7163.MCT-16-0205. Epub 2016 Nov 15. PMID 28062705

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 8 investigative sites in the United States and Canada from 08 Jun 2016 to 26 Jan 2021.
Pre-assignment Details: A total of 60 participants were enrolled and randomized to receive treatment in 2 phases, Dose Escalation (Part A [23 participants] and Part B [27 participants]; and Dose Expansion Phases (Part C [10 participants]). Study was terminated prematurely due to a lack of efficacy during primary analysis and therefore, efficacy, pharmacokinetic (PK) and pharmacodynamics (PDn) assessments were not determined.
Groups:
- Part A: KPT-9274 10mg: Participants received 10 milligrams (mg) of oral tablets of KPT-9274 three times a week every other day during each 28 day cycle.
- Part A: KPT-9274 20mg: Participants received 20mg of oral tablets of KPT-9274 three times a week every other day during each 28 day cycle.
- Part A: KPT-9274 30mg: Participants received 30mg of oral tablets of KPT-9274 three times a week every other day during each 28 day cycle.
- Part A: KPT-9274 40mg: Participants received 40mg of oral tablets of KPT-9274 three times a week every other day during each 28 day cycle.
Period: Overall Study
Arm/Group | Part A: KPT-9274 10mg | Part A: KPT-9274 20mg | Part A: KPT-9274 30mg | Part A: KPT-9274 40mg | Part A: KPT-9274 40mg BIW | Part B: KPT-9274 30mg + Niacin 500mg | Part B: KPT-9274 40mg + Niacin 500mg | Part B: KPT-9274 60mg + Niacin 500mg | Part B: KPT-9274 80mg + Niacin 500mg | Part B: KPT-9274 100mg + Niacin 500mg | Part C: KPT-9274 20mg + Nivolumab 480mg | Part C: KPT-9274 30mg + Nivolumab 480mg | Part C: KPT-9274 40mg + Nivolumab 480mg
Started | 3 | 3 | 5 | 7 | 5 | 3 | 4 | 12 | 7 | 1 | 1 | 5 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 5 | 7 | 5 | 3 | 4 | 12 | 7 | 1 | 1 | 5 | 4
Not completed — Disease progression | 3 | 3 | 2 | 4 | 4 | 1 | 2 | 8 | 5 | 1 | 0 | 3 | 2
Not completed — Clinical progression | 0 | 0 | 2 | 1 | 0 | 2 | 1 | 4 | 0 | 0 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population consisted of all participants who had received at least 1 dose of the study treatment. Participants were analyzed according to the treatment they received.
Groups:
- Part A: KPT-9274 10mg: Participants received 10mg of oral tablets of KPT-9274 three times a week every other day during each 28 day cycle.
- Part A: KPT-9274 40mg BIW: Participants received KPT-9274 40mg of oral tablet BIW during each 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Part A: KPT-9274 10mg | Part A: KPT-9274 20mg | Part A: KPT-9274 30mg | Part A: KPT-9274 40mg | Part A: KPT-9274 40mg BIW | Part B: KPT-9274 30mg + Niacin 500mg | Part B: KPT-9274 40mg + Niacin 500mg | Part B: KPT-9274 60mg + Niacin 500mg | Part B: KPT-9274 80mg + Niacin 500mg | Part B: KPT-9274 100mg + Niacin 500mg | Part C: KPT-9274 20mg + Nivolumab 480mg | Part C: KPT-9274 30mg + Nivolumab 480mg | Part C: KPT-9274 40mg + Nivolumab 480mg | Total
Number analyzed (Participants) | 3 | 3 | 5 | 7 | 5 | 3 | 4 | 12 | 7 | 1 | 1 | 5 | 4 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.3 (16.62) | 63.7 (3.21) | 56.6 (6.77) | 59.6 (17.17) | 68.8 (4.66) | 44.0 (14.73) | 65.0 (4.55) | 61.8 (9.69) | 55.0 (15.00) | 38.0 (NA) — Standard deviation was not calculated, as there is only one participant enrolled in this arm. | 67.0 (NA) — Standard deviation was not calculated, as there is only one participant enrolled in this arm. | 63.6 (14.36) | 62.0 (10.20) | 59.8 (12.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 2 | 1 | 1 | 3 | 6 | 2 | 0 | 0 | 5 | 2 | 26
  Male | 2 | 3 | 2 | 5 | 4 | 2 | 1 | 6 | 5 | 1 | 1 | 0 | 2 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 3 | 3 | 4 | 5 | 5 | 2 | 4 | 8 | 5 | 0 | 1 | 5 | 4 | 49
  Unknown or Not Reported | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 4
  White | 2 | 3 | 3 | 5 | 4 | 2 | 4 | 10 | 5 | 1 | 1 | 4 | 3 | 47
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) for KPT-9274
Description: The MTD was defined as the highest dose at which less than or equal to (<=) 1 participant experienced a dose limiting toxicity (DLT) in Cycle 1. A DLT was defined as an adverse event (AE) or abnormal laboratory value occurring within the first 28 days of treatment of KPT-9274, excluding those clearly caused by underlying disease, disease progression, or external factors.
Time Frame: From start of study drug administration up to 44 weeks
Population: Study was terminated prematurely due to a lack of efficacy. Therefore, the data were not determined due to insufficient number of participants with events.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: KPT-9274 10mg | Part A: KPT-9274 20mg | Part A: KPT-9274 30mg | Part A: KPT-9274 40mg | Part A: KPT-9274 40mg BIW | Part B: KPT-9274 30mg + Niacin 500mg | Part B: KPT-9274 40mg + Niacin 500mg | Part B: KPT-9274 60mg + Niacin 500mg | Part B: KPT-9274 80mg + Niacin 500mg | Part B: KPT-9274 100mg + Niacin 500mg | Part C: KPT-9274 20mg + Nivolumab 480mg | Part C: KPT-9274 30mg + Nivolumab 480mg | Part C: KPT-9274 40mg + Nivolumab 480mg
Number analyzed (Participants) | 3 | 3 | 5 | 7 | 5 | 3 | 4 | 12 | 7 | 1 | 1 | 5 | 4
Participants | NA — MTD was not determined based on insufficient number of participants with events. | NA — MTD was not determined based on insufficient number of participants with events. | NA — MTD was not determined based on insufficient number of participants with events. | NA — MTD was not determined based on insufficient number of participants with events. | NA — MTD was not determined based on insufficient number of participants with events. | NA — MTD was not determined based on insufficient number of participants with events. | NA — MTD was not determined based on insufficient number of participants with events. | NA — MTD was not determined based on insufficient number of participants with events. | NA — MTD was not determined based on insufficient number of participants with events. | NA — MTD was not determined based on insufficient number of participants with events. | NA — MTD was not determined based on insufficient number of participants with events. | NA — MTD was not determined based on insufficient number of participants with events. | NA — MTD was not determined based on insufficient number of participants with events.

2. Primary Outcome: Number of Dose Limiting Toxicities (DLT) Experienced by Participants
Description: A DLT was defined as an AE or abnormal laboratory value occurring within the first 28 days of KPT-9274 treatment, excluding those clearly caused by underlying disease, disease progression, or extraneous causes, and meets any of the criteria for defining dose limiting toxicities.
Time Frame: At Cycle 1 only (28-day cycle)
Population: The safety population consisted of all participants who had received at least 1 dose of the study treatment.
Measure: Number; unit: Number of DLTs
Arm/Group | Part A: KPT-9274 10mg | Part A: KPT-9274 20mg | Part A: KPT-9274 30mg | Part A: KPT-9274 40mg | Part A: KPT-9274 40mg BIW | Part B: KPT-9274 30mg + Niacin 500mg | Part B: KPT-9274 40mg + Niacin 500mg | Part B: KPT-9274 60mg + Niacin 500mg | Part B: KPT-9274 80mg + Niacin 500mg | Part B: KPT-9274 100mg + Niacin 500mg | Part C: KPT-9274 20mg + Nivolumab 480mg | Part C: KPT-9274 30mg + Nivolumab 480mg | Part C: KPT-9274 40mg + Nivolumab 480mg
Number analyzed (Participants) | 3 | 3 | 5 | 7 | 5 | 3 | 4 | 12 | 7 | 1 | 1 | 5 | 4
Number of DLTs | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Adverse Event (AE) of Severity Grade >= 3 or 4, Serious AEs, and AEs Leading to Treatment Discontinuation
Description: The AE severity was graded on a scale from 1 to 4 using the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.03; any events not specifically listed in the scale were defined as: Grade 1 is mild; Grade 2 is moderate; Grade 3 is severe or medically significant; Grade 4 is life-threatening. An SAE was any untoward medical occurrence that at any dose met one, more of the following criteria: results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent, significant disability/incapacity, a congenital abnormality/birth defect, an important medical event. The AE leading to treatment discontinuation in the study.
Time Frame: From start of study drug administration up to 49 weeks
Population: The safety population consisted of all participants who had received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: KPT-9274 10mg | Part A: KPT-9274 20mg | Part A: KPT-9274 30mg | Part A: KPT-9274 40mg | Part A: KPT-9274 40mg BIW | Part B: KPT-9274 30mg + Niacin 500mg | Part B: KPT-9274 40mg + Niacin 500mg | Part B: KPT-9274 60mg + Niacin 500mg | Part B: KPT-9274 80mg + Niacin 500mg | Part B: KPT-9274 100mg + Niacin 500mg | Part C: KPT-9274 20mg + Nivolumab 480mg | Part C: KPT-9274 30mg + Nivolumab 480mg | Part C: KPT-9274 40mg + Nivolumab 480mg
Number analyzed (Participants) | 3 | 3 | 5 | 7 | 5 | 3 | 4 | 12 | 7 | 1 | 1 | 5 | 4
Participants
  Maximum Grade 3/4 AEs | 1 | 2 | 5 | 7 | 3 | 2 | 3 | 10 | 7 | 1 | 1 | 4 | 3
  Maximum Grade 4 AEs | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Serious AEs | 0 | 2 | 2 | 3 | 0 | 1 | 1 | 6 | 1 | 1 | 1 | 2 | 2
  AEs Leading to Study Treatment Discontinuation | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1

4. Primary Outcome: Percentage of Participants With Overall Response Rate (ORR)
Description: The ORR was defined as percentage of participants who had a response of partial response (PR) or complete response (CR). The PR was achieved when a participant had at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. The CR was achieved in a participant when all target lesions disappeared. Any pathological lymph nodes (whether target or non target) must have reduction in the short axis to <10 millimeter (mm).
Time Frame: From date of randomization up to 44 weeks
Population: Study was terminated prematurely due to a lack of efficacy during primary analysis stage. Data for this outcome measure was not collected or analyzed as per planned analysis.
Arm/Group | Part A: KPT-9274 10mg | Part A: KPT-9274 20mg | Part A: KPT-9274 30mg | Part A: KPT-9274 40mg | Part A: KPT-9274 40mg BIW | Part B: KPT-9274 30mg + Niacin 500mg | Part B: KPT-9274 40mg + Niacin 500mg | Part B: KPT-9274 60mg + Niacin 500mg | Part B: KPT-9274 80mg + Niacin 500mg | Part B: KPT-9274 100mg + Niacin 500mg | Part C: KPT-9274 20mg + Nivolumab 480mg | Part C: KPT-9274 30mg + Nivolumab 480mg | Part C: KPT-9274 40mg + Nivolumab 480mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Percentage of Participants With Disease Control Rate (DCR)
Description: The DCR was defined as percentage of participants who have a response of CR, PR, and stable disease (SD) >= 16 weeks, DCR = CR + PR+ SD. The PR was achieved when a participant had at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. The CR was achieved in a participant when all target lesions disappeared. Any pathological lymph nodes (whether target or non-target) must have reduction in the short axis to <10mm. The SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD).
Time Frame: From date of the first study treatment up to 44 weeks
Population: as for outcome 4
Arm/Group | Part A: KPT-9274 10mg | Part A: KPT-9274 20mg | Part A: KPT-9274 30mg | Part A: KPT-9274 40mg | Part A: KPT-9274 40mg BIW | Part B: KPT-9274 30mg + Niacin 500mg | Part B: KPT-9274 40mg + Niacin 500mg | Part B: KPT-9274 60mg + Niacin 500mg | Part B: KPT-9274 80mg + Niacin 500mg | Part B: KPT-9274 100mg + Niacin 500mg | Part C: KPT-9274 20mg + Nivolumab 480mg | Part C: KPT-9274 30mg + Nivolumab 480mg | Part C: KPT-9274 40mg + Nivolumab 480mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Progression-free Survival (PFS)
Description: The PFS was defined as the duration of time from date of the first study treatment until the first date that PD is objectively documented or death due to any cause. The PD is defined as at least a 20% increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded since the treatment started. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. Appearance of one or more new lesions will also constitute PD.
Time Frame: From the date of first study treatment until the first date of PD, or death due (up to 44 weeks)
Population: as for outcome 4
Arm/Group | Part A: KPT-9274 10mg | Part A: KPT-9274 20mg | Part A: KPT-9274 30mg | Part A: KPT-9274 40mg | Part A: KPT-9274 40mg BIW | Part B: KPT-9274 30mg + Niacin 500mg | Part B: KPT-9274 40mg + Niacin 500mg | Part B: KPT-9274 60mg + Niacin 500mg | Part B: KPT-9274 80mg + Niacin 500mg | Part B: KPT-9274 100mg + Niacin 500mg | Part C: KPT-9274 20mg + Nivolumab 480mg | Part C: KPT-9274 30mg + Nivolumab 480mg | Part C: KPT-9274 40mg + Nivolumab 480mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Overall Survival (OS)
Description: The OS was defined as the duration of time from date of the first study treatment until death from any cause.
Time Frame: From date of the first study treatment until death (up to 44 weeks)
Population: as for outcome 4
Arm/Group | Part A: KPT-9274 10mg | Part A: KPT-9274 20mg | Part A: KPT-9274 30mg | Part A: KPT-9274 40mg | Part A: KPT-9274 40mg BIW | Part B: KPT-9274 30mg + Niacin 500mg | Part B: KPT-9274 40mg + Niacin 500mg | Part B: KPT-9274 60mg + Niacin 500mg | Part B: KPT-9274 80mg + Niacin 500mg | Part B: KPT-9274 100mg + Niacin 500mg | Part C: KPT-9274 20mg + Nivolumab 480mg | Part C: KPT-9274 30mg + Nivolumab 480mg | Part C: KPT-9274 40mg + Nivolumab 480mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Time to Progression (TTP)
Description: The TTP was defined as the duration of time from date of the first study treatment until the first date that PD was objectively documented or death due to PD.
Time Frame: From date of the first study treatment until the first date of PD or death (up to 44 weeks)
Population: as for outcome 4
Arm/Group | Part A: KPT-9274 10mg | Part A: KPT-9274 20mg | Part A: KPT-9274 30mg | Part A: KPT-9274 40mg | Part A: KPT-9274 40mg BIW | Part B: KPT-9274 30mg + Niacin 500mg | Part B: KPT-9274 40mg + Niacin 500mg | Part B: KPT-9274 60mg + Niacin 500mg | Part B: KPT-9274 80mg + Niacin 500mg | Part B: KPT-9274 100mg + Niacin 500mg | Part C: KPT-9274 20mg + Nivolumab 480mg | Part C: KPT-9274 30mg + Nivolumab 480mg | Part C: KPT-9274 40mg + Nivolumab 480mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Duration of Response (DOR)
Description: The DOR was defined as the duration of time from the first meeting CR or PR measurement criteria (whichever occurs first) until the first date diseases progression.
Time Frame: Up to 44 weeks
Population: as for outcome 4
Arm/Group | Part A: KPT-9274 10mg | Part A: KPT-9274 20mg | Part A: KPT-9274 30mg | Part A: KPT-9274 40mg | Part A: KPT-9274 40mg BIW | Part B: KPT-9274 30mg + Niacin 500mg | Part B: KPT-9274 40mg + Niacin 500mg | Part B: KPT-9274 60mg + Niacin 500mg | Part B: KPT-9274 80mg + Niacin 500mg | Part B: KPT-9274 100mg + Niacin 500mg | Part C: KPT-9274 20mg + Nivolumab 480mg | Part C: KPT-9274 30mg + Nivolumab 480mg | Part C: KPT-9274 40mg + Nivolumab 480mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Maximum Plasma Concentration (Cmax) in Participants Who Received KPT-9274
Description: Cmax achieved by the KPT-9274 after the first dose administrations.
Time Frame: Cycle 1 and 2: Pre-dose, 3, 6, 8, 24, and 48 hours post-dose (each cycle =28 days)
Population: as for outcome 4
Groups:
- Part A: KPT-9274 40mg BIW: Participants received KPT-9274 20mg of oral tablet biweekly (BIW) during each 28-day cycle.
Arm/Group | Part A: KPT-9274 10mg | Part A: KPT-9274 20mg | Part A: KPT-9274 30mg | Part A: KPT-9274 40mg | Part A: KPT-9274 40mg BIW | Part B: KPT-9274 30mg + Niacin 500mg | Part B: KPT-9274 40mg + Niacin 500mg | Part B: KPT-9274 60mg + Niacin 500mg | Part B: KPT-9274 80mg + Niacin 500mg | Part B: KPT-9274 100mg + Niacin 500mg | Part C: KPT-9274 20mg + Nivolumab 480mg | Part C: KPT-9274 30mg + Nivolumab 480mg | Part C: KPT-9274 40mg + Nivolumab 480mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Time-to-peak Plasma Concentration (Tmax) in Participants Who Received KPT-9274
Description: Time taken by KPT-9274 to achieve maximum plasma concentration after the first dose administration.
Time Frame: Cycle 1 and 2: Pre-dose, 3, 6, 8, 24, and 48 hours post-dose (each cycle =28 days)
Population: as for outcome 4
Arm/Group | Part A: KPT-9274 10mg | Part A: KPT-9274 20mg | Part A: KPT-9274 30mg | Part A: KPT-9274 40mg | Part A: KPT-9274 40mg BIW | Part B: KPT-9274 30mg + Niacin 500mg | Part B: KPT-9274 40mg + Niacin 500mg | Part B: KPT-9274 60mg + Niacin 500mg | Part B: KPT-9274 80mg + Niacin 500mg | Part B: KPT-9274 100mg + Niacin 500mg | Part C: KPT-9274 20mg + Nivolumab 480mg | Part C: KPT-9274 30mg + Nivolumab 480mg | Part C: KPT-9274 40mg + Nivolumab 480mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Terminal Half-life (T1/2) in Participants Who Received KPT-9274
Description: The T1/2 was defied as the time it takes for the concentration of KPT-9274 in the plasma to be reduced by 50%.
Time Frame: Cycle 1 and 2: Pre-dose, 3, 6, 8, 24, and 48 hours post-dose (each cycle =28 days)
Population: as for outcome 4
Arm/Group | Part A: KPT-9274 10mg | Part A: KPT-9274 20mg | Part A: KPT-9274 30mg | Part A: KPT-9274 40mg | Part A: KPT-9274 40mg BIW | Part B: KPT-9274 30mg + Niacin 500mg | Part B: KPT-9274 40mg + Niacin 500mg | Part B: KPT-9274 60mg + Niacin 500mg | Part B: KPT-9274 80mg + Niacin 500mg | Part B: KPT-9274 100mg + Niacin 500mg | Part C: KPT-9274 20mg + Nivolumab 480mg | Part C: KPT-9274 30mg + Nivolumab 480mg | Part C: KPT-9274 40mg + Nivolumab 480mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Volume of Distribution (Vd/F) in Participants Who Received KPT-9274
Description: The Vd/F was defined as MRT*CL/F, where MRT is the mean residence time (calculated as AUMC[0-tau]/AUC[0-tau], where AUMC[0-tau] is the area under the first moment curve determined as the area under the concentration*time versus time curve).
Time Frame: Cycle 1 and 2: Pre-dose, 3, 6, 8, 24, and 48 hours post-dose (each cycle =28 days)
Population: as for outcome 4
Arm/Group | Part A: KPT-9274 10mg | Part A: KPT-9274 20mg | Part A: KPT-9274 30mg | Part A: KPT-9274 40mg | Part A: KPT-9274 40mg BIW | Part B: KPT-9274 30mg + Niacin 500mg | Part B: KPT-9274 40mg + Niacin 500mg | Part B: KPT-9274 60mg + Niacin 500mg | Part B: KPT-9274 80mg + Niacin 500mg | Part B: KPT-9274 100mg + Niacin 500mg | Part C: KPT-9274 20mg + Nivolumab 480mg | Part C: KPT-9274 30mg + Nivolumab 480mg | Part C: KPT-9274 40mg + Nivolumab 480mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Apparent Plasma Clearance (CL/F) in Participants Who Received KPT-9274
Description: The CL/F was calculated as the KPT-9274 dose administered divided by the area-under-the-curve of KPT-9274 plasma concentration versus (vs) time.
Time Frame: Cycle 1 and 2: Pre-dose, 3, 6, 8, 24, and 48 hours post-dose (each cycle =28 days)
Population: as for outcome 4
Arm/Group | Part A: KPT-9274 10mg | Part A: KPT-9274 20mg | Part A: KPT-9274 30mg | Part A: KPT-9274 40mg | Part A: KPT-9274 40mg BIW | Part B: KPT-9274 30mg + Niacin 500mg | Part B: KPT-9274 40mg + Niacin 500mg | Part B: KPT-9274 60mg + Niacin 500mg | Part B: KPT-9274 80mg + Niacin 500mg | Part B: KPT-9274 100mg + Niacin 500mg | Part C: KPT-9274 20mg + Nivolumab 480mg | Part C: KPT-9274 30mg + Nivolumab 480mg | Part C: KPT-9274 40mg + Nivolumab 480mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 49 weeks
Groups:
- Part B: KPT-9274 30mg + Niacin 500mg: Participants received KPT-9274 30mg of oral tablet along with a starting dose of 500mg niacin ER orally three times a week every other day during each 28-day cycle.
- Experimental: Part B: KPT-9274 100mg + Niacin 500mg: Participants received KPT-9274 100mg of oral tablet along with a starting dose of 500mg niacin ER orally three times a week every other day during each 28-day cycle.
Arm/Group | Part A: KPT-9274 10mg | Part A: KPT-9274 20mg | Part A: KPT-9274 30mg | Part A: KPT-9274 40mg | Part A: KPT-9274 40mg BIW | Part B: KPT-9274 30mg + Niacin 500mg | Part B: KPT-9274 40mg + Niacin 500mg | Part B: KPT-9274 60mg + Niacin 500mg | Part B: KPT-9274 80mg + Niacin 500mg | Experimental: Part B: KPT-9274 100mg + Niacin 500mg | Part C: KPT-9274 20mg + Nivolumab 480mg | Part C: KPT-9274 30mg + Nivolumab 480mg | Part C: KPT-9274 40mg + Nivolumab 480mg
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/3 | 3/5 | 5/7 | 1/5 | 3/3 | 3/4 | 6/12 | 4/7 | 1/1 | 1/1 | 2/5 | 3/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/3 | 2/5 | 3/7 | 0/5 | 1/3 | 1/4 | 6/12 | 1/7 | 1/1 | 1/1 | 2/5 | 2/4
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 5/5 | 7/7 | 5/5 | 3/3 | 4/4 | 12/12 | 7/7 | 1/1 | 1/1 | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: KPT-9274 10mg (N=3) | Part A: KPT-9274 20mg (N=3) | Part A: KPT-9274 30mg (N=5) | Part A: KPT-9274 40mg (N=7) | Part A: KPT-9274 40mg BIW (N=5) | Part B: KPT-9274 30mg + Niacin 500mg (N=3) | Part B: KPT-9274 40mg + Niacin 500mg (N=4) | Part B: KPT-9274 60mg + Niacin 500mg (N=12) | Part B: KPT-9274 80mg + Niacin 500mg (N=7) | Experimental: Part B: KPT-9274 100mg + Niacin 500mg (N=1) | Part C: KPT-9274 20mg + Nivolumab 480mg (N=1) | Part C: KPT-9274 30mg + Nivolumab 480mg (N=5) | Part C: KPT-9274 40mg + Nivolumab 480mg (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intracranial mass (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: KPT-9274 10mg (N=3) | Part A: KPT-9274 20mg (N=3) | Part A: KPT-9274 30mg (N=5) | Part A: KPT-9274 40mg (N=7) | Part A: KPT-9274 40mg BIW (N=5) | Part B: KPT-9274 30mg + Niacin 500mg (N=3) | Part B: KPT-9274 40mg + Niacin 500mg (N=4) | Part B: KPT-9274 60mg + Niacin 500mg (N=12) | Part B: KPT-9274 80mg + Niacin 500mg (N=7) | Experimental: Part B: KPT-9274 100mg + Niacin 500mg (N=1) | Part C: KPT-9274 20mg + Nivolumab 480mg (N=1) | Part C: KPT-9274 30mg + Nivolumab 480mg (N=5) | Part C: KPT-9274 40mg + Nivolumab 480mg (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 5 | 7 | 5 | 1 | 2 | 8 | 7 | 1 | 1 | 5 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 3 | 2 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 5 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 3 | 1 | 3 | 6 | 5 | 1 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 3 | 4 | 3 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 2 | 4 | 2 | 2 | 2 | 4 | 5 | 0 | 0 | 2 | 2
Oedema peripheral (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 2 | 1 | 1 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 5 | 2 | 2 | 1 | 2 | 1 | 1 | 0 | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3 | 0 | 1 | 0 | 3 | 4 | 1 | 1 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pupils unequal (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Blood iron decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Reticulocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 5 | 2 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 4 | 2 | 1 | 0 | 3 | 2 | 1 | 0 | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin B12 decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glucose urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Generalised oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Study was terminated prematurely due to a lack of efficacy during primary analysis and therefore, efficacy, PK and PDn assessments were not determined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT02702492/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT02702492/SAP_001.pdf